CLINICAL TRIAL: NCT00307060
Title: A Randomized, Double-Blind, Parallel-Filter Study to Evaluate the Antihypertensive Efficacy and Safety of Losartan-HCTZ Combination as Compared to Losartan Monotherapy in Patients With Essential Hypertension
Brief Title: MK0954A-264 Filter Study (0954A-264)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0954A-264; 2006_019
Record Dates: First submitted 2006-03-23; First posted 2006-03-27 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Mild to Severe Hypertension
MeSH Terms: interventions — Hydrochlorothiazide; Losartan; Duration of Therapy

INTERVENTIONS:
Drug: MK0954A, hydrochlorothiazide (+) losartan potassium / Duration of Treatment: 6 weeks
Drug: losartan / Duration of Treatment: 6 weeks

SUMMARY:
To compare the blood pressure lowering efficacy, safety and tolerability of a combination drug to a single drug taken once daily in patients with uncontrolled blood pressure following a 4-week filter on the single therapy product.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with mild to severe hypertension (SiDBP 90-120 mmHg)

Exclusion Criteria:

* Systolic BP > 200 mmHg
* Secondary or malignant hypertension
* Taking more than 2 antihypertensive medications
* Hypertension induced by oral contraceptives
* Hx of cerebral vascular accident within 6 months
* Hx of angina, myocardial infarction, PCI, CABG, or decompensated CHF within 6 months
* Clinically significant AV conduction disturbance or potentially life threatening ventricular arrhythmias, valvular disease, cardiomyopathy, unexplained syncope
* History of angioedema
* Sensitivity to AII receptor antagonists or HCTZ, nephrotic syndrome,single kidney function
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2004-12-01 (Actual); Primary Completion 2005-06-01 (Actual); Study Completion 2005-06-02 (Actual)

PRIMARY OUTCOMES:
Losartan-HCTZ 100-12.5 mg combination will be more effective in lower mean through sitting diastolic blood pressure (SiDBP) than losartan 100 mg monotherapy after 6 weeks of treatment. | 6 Weeks

SECONDARY OUTCOMES:
Losartan-HCTZ 100-12.5 mg combination will be more effective in lowering mean through sitting systolic blood pressure (SiSBP) after 6 weeks of treatment compared to losartan 100-mg monotherapy, and will be safe and tolerable. | 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Gleim GW, Rubino J, Zhang H, Shahinfar S, Soffer BA, Lyle PA, Littlejohn TW 3rd, Feig PU. A multicenter, randomized, double-blind, parallel-group trial of the antihypertensive efficacy and tolerability of a combination of once-daily losartan 100 mg/hydrochlorothiazide 12.5 mg compared with losartan 100-mg monotherapy in the treatment of mild to severe essential hypertension. Clin Ther. 2006 Oct;28(10):1639-48. doi: 10.1016/j.clinthera.2006.10.014. PMID 17157119